CLINICAL TRIAL: NCT01745328
Title: Study on Treatment of Recurrent Urinary Tract Infection by Traditional Chinese Medicine
Brief Title: Treatment of Recurrent Urinary Tract Infection (RUTI) by Traditional Chinese Medicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Institute of Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WJUTI
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: recurrent urinary tract infection; antibiotics; traditional chinese medicine
MeSH Terms: conditions — Urinary Tract Infections | interventions — Levofloxacin; BID protein, human; Amoxicillin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LVX-AMX (Active Comparator): subject is treated with LAV-AMX, then followed by placebo.
  Interventions: Drug: LVX-AMX
- TCM treatment (Active Comparator): subject is treated with TCM
  Interventions: Drug: TCM

INTERVENTIONS:
Drug: LVX-AMX — Subjects were treated with Levofloxacin, 200mg bid, Amoxicillin, 500mg tid for 1 week, followed by 3 week of placebo.
  Other Names: Levofloxacin, 200mg bid, Amoxicillin, 500mg tid
  Arms: LVX-AMX
Drug: TCM — Subject is treated with TCM for 4 weeks.
  Other Names: TCM formula consisted of 10 herbals
  Arms: TCM treatment
Drug: LVX-AMX — treatment with placebo from 2 to 4 weeks.
  Other Names: placebo from 2 to 4 weeks.
  Arms: LVX-AMX

SUMMARY:
Traditional Chinese Medicine (TCM) could be used to treat Recurrent urinary tract infection (RUTI).

DETAILED DESCRIPTION:
Antibiotics and TCM are used to treat RUTI to evaluate treatment efficiencies.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated RUTI

Exclusion Criteria:

* complicated RUTI
* other disease with urinary tract
* infection by pathogens other than bacteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Recovery of recurrent urinary tract infection | 4 weeks after study drug start
  Patients are checked at 4 weeks at the end of the treatment to confirm recovery of RUTI.

SECONDARY OUTCOMES:
Urinary albumin | 4 weeks after drug start
  Urinary albumin is checked in patient urine.
WBC conversion | 4 weeks after drug start
  Check the WBC count in patient urine.
Urination frequency | 4 weeks after drug start
  Checked for urination frequency at 4 weeks after drug start.
Recurrence | 6 months after drug start
  Patients are checked for recurrence rate at 6 months after drug start by telephone interview.
urgency | 4 weeks after drug start
  Check urgency 4 weeks after drug start

CONTACTS AND LOCATIONS:
Overall Officials: Zeliang Chen, Dr, Principal Investigator — Insititute of Disease Control and Prevention
Locations (1):
- Wangjing Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu SW, Guo J, Wu WK, Chen ZL, Zhang N. Treatment of Uncomplicated Recurrent Urinary Tract Infection with Chinese Medicine Formula: A Randomized Controlled Trial. Chin J Integr Med. 2019 Jan;25(1):16-22. doi: 10.1007/s11655-017-2960-4. Epub 2017 Jul 25. PMID 28741061